CLINICAL TRIAL: NCT01579383
Title: A Single Dose, Placebo-Controlled, Ascending Dose Study to Determine the Safety, Tolerability and Pharmacokinetics of ALD403, a Humanized Anti-Calcitonin Gene-Related Peptide Monoclonal Antibody Administered by Intravenous Infusion and Subcutaneous Injection
Brief Title: Safety Tolerability and Pharmacokinetics of ALD403
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ALD403-CLIN-001
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Migraine Disorders
Keywords: Migraine Disorders; Phase 1; ALD403
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A, Cohorts A - H (Experimental): ALD403/Placebo
  Interventions: Biological: ALD403
- Part A, Cohort I (Experimental): ALD403/Placebo
  Interventions: Biological: ALD403
- Part B (Experimental): ALD403/Placebo/Sumatriptan
  Interventions: Biological: ALD403; Biological: Sumatriptan

INTERVENTIONS:
Biological: ALD403 — Single Dose IV infusion on Day 1
  Arms: Part A, Cohorts A - H; Part B
Biological: ALD403 — Single Dose subcutaneous injection on Day 1
  Arms: Part A, Cohort I
Biological: Sumatriptan — Single Dose subcutaneous injection on Day 1
  Arms: Part B

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of ALD403, a monoclonal antibody, administered by intravenous infusion and subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria Part A:

* Healthy males and females between the ages of 18 and 65 (inclusive).
* Normal renal function as calculated by the Cockcroft- Gault equation at screening.
* Body Mass Index (BMI) between 18.0 and 30.0 kg/m2, and a total body weight of 50 to 100kg inclusive.
* No clinically significant disease or abnormal laboratory values as determined by medical history, physical examination, electrocardiogram, and laboratory evaluations

Exclusion Criteria Part A:

* History of febrile illness within 5 days prior to the first dose
* Any clinically significant laboratory findings
* Any clinically significant physical exam abnormalities
* Hospitalization for any reason within 30 days of the screening visit.
* History of or positive human immunodeficiency virus (HIV) screen result
* History of positive Hepatitis B surface antigen (HBsAg), and/or positive Hepatitis C antibody (HCV) at screening.
* History of malignancy within five years prior to screening.
* History of leukemia, myeloproliferative disorder or lymphoproliferative disorder
* History of rubber, latex allergy or allergy to medical adhesives
* Positive urine, drug or alcohol screen result
* Current smokers
* Previous treatment or clinical trial with a monoclonal antibody.
* Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives

Inclusion Criteria Part B:

* Healthy females between the ages of 18 and 65 (inclusive).
* Male and female migraine patients with clinically diagnosed migraine not attributed to another cause with or without aura based on International Headache Society criteria.
* Migraine patients must have a history of migraine with or without aura for more than 1 year with 1-8 moderate or severe migraine attacks per month in the 2 months prior to starting in the study.
* Normal renal function as defined by Cockcroft- Gault equation at screening.
* Body Mass Index (BMI) between 18.0 and 30.0 kg/m2, and a total body weight of 50 to 100kg inclusive.
* No clinically significant disease or abnormal laboratory values as determined by medical history, physical examination, electrocardiogram, and laboratory evaluations conducted at the screening visit or at the time of admission

Exclusion Criteria Part B:

* For migraine patients: patient is not able to refrain from use of their usual triptan therapy (if applicable) from 48 hours (Day -2) prior to dosing on Day 1 until the morning of discharge (Day 3).
* Migraine patients who experience migraine with prolonged aura, familiar hemiplegic migraine, migrainous infarction or basilar migraine
* For migraine patients: patient has more than 8 headache-days per month or has taken medication for acute headache on more than 8 days a month in the past 3 months
* For migraine patients: patient was greater than 50 years old at the age of migraine onset
* History of febrile illness within 5 days prior to the first dose
* Any clinically significant laboratory findings
* Any clinically significant physical exam abnormalities
* Previous treatment or clinical trial with a monoclonal antibody.
* Hospitalization for any reason within 30 days of the screening visit.
* History of or positive human immunodeficiency virus (HIV) screen result
* History of positive Hepatitis B surface antigen (HBsAg), and/or positive Hepatitis C antibody (HCV
* History of malignancy within five years prior to screening.
* History of leukemia, myeloproliferative disorder or lymphoproliferative disorder
* Positive urine drug or alcohol screen result
* Current smokers.
* Known contraindication to sumatriptan
* Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ALD403: laboratory variables, ECG and adverse events | 12 weeks
  * Physical Examination
  * Vital signs
  * 12-lead ECG (electrocardiogram)
  * Clinical laboratory tests (hematology, chemistry)
  * Number of participants with Adverse Events

SECONDARY OUTCOMES:
Evaluation of Pharmacokinetics of ALD403 | 12 weeks
  * Cmax - maximum plasma concentration
  * Tmax - Time to achieve maximum plasma concentration
  * AUC - Area under the plasma concentration-time curve
  * T1/2 - Elimination half-life
  * Vz - Volume of distribution
  * CL - Clearance
  * Bioavailability
Evaluation of pharmacodynamics of ALD403 | 12 weeks
  * Blood perfusion rates
  * Plasma levels of unbound ALD403
  * Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hodsman, MD, Principal Investigator — Nucleus Network
Locations (1):
- Centre for Clinical Studies, Nucleus Network, Melbourne, Victoria, Australia